CLINICAL TRIAL: NCT03084952
Title: A Phase 2, Randomized, Unicentric Clinical Trial With Dose Scaling for Safety, Tolerability and Efficacy Assessment of 18-Methoxycoronaridine Administered to Cutaneous Leishmaniasis Patients
Brief Title: Phase 2 Trial to Evaluate 18-Methoxycoronaridine Efficacy, Safety and Tolerability in Cutaneous Leishmaniasis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Infan Industria Quimica Farmaceutica Nacional (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB/F2-002/2016
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Leishmaniasis; American, Cutaneous; Drug Side Effect
Keywords: safety; pharmacokynetics; leishmaniasis treatment
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Drug-Related Side Effects and Adverse Reactions | interventions — 18-methoxycoronaridine; Meglumine Antimoniate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1 mg/day (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine
- 4 mg/day (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine
- 8 mg/day (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine
- 12 mg/day (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine
- Glucantime (Active Comparator)
  Interventions: Drug: Glucantime
- Best dose 18-MC (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine
- Minimum effective dose 18-MC (Experimental)
  Interventions: Drug: 18-Methoxycoronaridine

INTERVENTIONS:
Drug: 18-Methoxycoronaridine — Drug under evaluation for leishmaniasis treatment
  Arms: 1 mg/day; 12 mg/day; 4 mg/day; 8 mg/day; Best dose 18-MC; Minimum effective dose 18-MC
Drug: Glucantime — Leishmaniasis standard drug in Brazil
  Arms: Glucantime

SUMMARY:
It is a randomized phase II clinical study, unicentre aimed to evaluate the tolerability, safety and efficacy of 18-Methoxyoronaridine as a candidate of tegumentary leishmaniasis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 59 years of age;
* Clinical diagnosis of leishmaniasis with at least one ulcerated lesion with evolution time from one month;
* Parasitological confirmation;
* Women of childbearing potential should not be pregnant or breastfeeding, confirmed by examination of b-HCG (Gonadotrophic-Chorionic Hormone beta) at the time of screening;
* Men and women should use barrier contraceptive methods during the course of the study;

Exclusion Criteria:

* History of any disease or comorbidities that, in the opinion of the investigator, can either put the individual at risk or influence the results and ability of the subject to participate in the study;
* History or presence of gastrointestinal, hepatic, cardiac, renal disease or any other known condition that may interfere with the absorption, distribution, metabolism or excretion of the investigational product;
* Any evidence of underlying serious disease (cardiac, renal, hepatic or pulmonary);
* Pregnancy or the patient's unwillingness to use barrier contraceptive methods during and 3 months after therapy;
* History of gastrointestinal ulcer disease, inflammatory bowel disease, symptoms of indigestion;
* Any clinically important abnormality in biochemistry, hematology, urinalysis or clinical outcomes judged by the investigator;
* Any positive screening result for hepatitis B antigens, hepatitis C antibodies, and human immunodeficiency virus (HIV);
* Any clinically significant abnormalities in the rate, or driving the resting ECG morphology that may interfere with the interpretation of the QT interval variations;
* History of cancer;
* History of drug abuse, judging by the investigator
* History of alcohol abuse or excessive alcohol consumption, judged by the investigator;
* History of smoking
* History of severe allergy / hypersensitivity, judged by the investigator;
* History of hypersensitivity to drugs with similar chemical structure.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Lesion Reduction and Re-epithelization - Definitive Cure | 6 months at the follow-up visit.
  complete epithelization of all ulcers and complete disappearance of inflammatory hardening of all lesions at 6 months at the follow-up visit.
Lesion Reduction and Re-epithelization - Partial Cure | 6 months at the follow-up visit.
  incomplete epithelialization or incomplete regression of inflammatory hardening of one or more lesions, and without the appearance of new lesions.
  Apparent cure: complete epithelization of all ulcers and regression ≥ 70% of the inflammatory hardening of all lesions.
Clinical Failure | 6 months at the follow-up visit.
  Any of the following topics as clinical failure: residual readers with the presence of non-GiemsaDiff-Quick print parasites, or the appearance of new lesions or ≥ 20% increase or no improvement of lesions previously documented.

IPD SHARING:
Plan to Share IPD: Undecided